CLINICAL TRIAL: NCT04114357
Title: Evaluating the Effect of Prebiotics on the Gut Microbiome Profile and Beta Cell Function in Newly Diagnosed Type 1 Diabetes
Brief Title: Effect of Prebiotics on the Gut Microbiome Profile and Beta Cell Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Heba M. Ismail, Assistant Professor of Pediatrics, Indiana University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1907172784; KL2TR002530 (NIH); UL1TR002529 (NIH)
Record Dates: First submitted 2019-09-30; First posted 2019-10-03 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Supplement Intervention and Control Diet, then Control Diet Alone (Experimental): This group will first consume the supplement daily for 4 weeks in addition to the diabetic diet then cross-over to follow the diabetic diet for 4 weeks.
  Interventions: Drug: Acetylated and Butyrylated High Amylose Maize Starch
- Control Diet Alone, then Supplement Intervention and Control Diet (No Intervention): This group will follow the control diet for 4 weeks first then cross-over to receive the supplement for 4 weeks in addition to the diabetic diet.

INTERVENTIONS:
Drug: Acetylated and Butyrylated High Amylose Maize Starch — Participants will be instructed to consume HAMS-AB in two divided doses at breakfast and dinner for 4 weeks
  Other Names: Hylon™ VII Butyrate, Hylon™ VII Acetate
  Arms: Supplement Intervention and Control Diet, then Control Diet Alone

SUMMARY:
Data suggest that intestinal microbiota might be critically involved both in autoimmunity and in glucose homeostasis. An acetylated and butyrylated form of high amylose maize starch (HAMS-AB) that increases beneficial short chain fatty acid (SCFA) production has been safe and effective in disease prevention in mouse type 1 diabetes (T1D) models. The objective of this application is to assess the effect of administering a prebiotic, such as HAMS- AB, on the gut microbiome profile, glycemia and β-cell function in humans with T1D.

DETAILED DESCRIPTION:
This is a pilot, single center clinical trial to evaluate the effect of using the prebiotic, HAMS-AB, on the gut microbiome profile, glycemia and β-cell function in children and adolescents ages 12-16 years with recently diagnosed type 1 diabetes.

Approximately 12 participants will be randomized to first to take the supplement and follow the diabetic diet or follow a diabetic diet alone for 4 weeks and then cross-over after a 4 week washout period.

The primary objective is to determine the effect of using the prebiotic on the gut microbiome profile in youth with T1D.

The secondary objectives are to determine the effect of using the prebiotic on SCFA production, glycemia and β-cell health and function.

Exploratory outcomes include changes in MAIT cells.

ELIGIBILITY:
Inclusion Criteria:

* Be between 11-17 years of age
* Willing to consume HAMS-AB and follow a diabetic diet
* Diagnosed by American Diabetes Association criteria with T1D in the last 4-36 months
* Random non-fasting C-peptide of 0.17nmol/ml or greater
* Willing to use an effective form of contraception if sexually active
* BMI< 85% for age and sex
* Positive for any one of the following diabetes-related autoantibodies that are tested clinically [insulin autoantibody (if tested within 14 days of diagnosis), glutamic acid decarboxylase (GAD), insulinoma-associated protein-2 (IA-2), or Zinc transporter 8 autoantibodies (ZnT8)].

Exclusion Criteria:

1. Presence of severe, active disease that interferes with dietary intake or requires the use of chronic medication, except for well-controlled hypothyroidism and mild asthma not requiring oral steroids.
2. Diabetes other than T1D (Known monogenic forms of diabetes, Type 2 diabetes)
3. Chronic illness known to affect glucose metabolism (e.g. Cushing syndrome, polycystic ovarian disorder, cystic fibrosis) or taking medications that affect glucose metabolism (e.g. steroids, metformin)
4. Psychiatric impairment or current use of anti-psychotic medication
5. Any condition that, in the investigator's opinion, may compromise study participation or may confound the interpretation of the study results.
6. Female participants of child-bearing age with reproductive potential, must not be pregnant and agree to use an effective form of birth control or be abstinent during the study period (see below)
7. History of recurrent infections
8. History of on-going infections or antibiotic treatment within the past three months
9. History of immune compromise
10. Steroid intake (inhaled or oral)
11. Other immunosuppressant use in past 6 months
12. History of gastrointestinal disease
13. Possible or confirmed celiac disease
14. Pregnancy or possible pregnancy
15. Allergy to corn (prebiotic)
16. Allergy to milk or milk products or soy present in Boost
17. Participation in other intervention research trials within the past 3 months
18. Anticipate major changes in diabetes management during study (change from injection to pump, new start of continuous glucose monitoring)
19. Consuming high fiber or vegetarian diet (consuming three or more servings of high fiber foods on 4 or more days per week) using validated dietary assessments (see below under schedule of events table).
20. Taking fiber supplements

    -

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-06-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ismail HM, Spall M, Evans-Molina C, DiMeglio LA. Evaluating the effect of prebiotics on the gut microbiome profile and beta cell function in youth with newly diagnosed type 1 diabetes: protocol of a pilot randomized controlled trial. Pilot Feasibility Stud. 2023 Aug 25;9(1):150. doi: 10.1186/s40814-023-01373-4. PMID 37626387

RESULTS

PARTICIPANT FLOW:
Groups:
- Supplement Intervention and Control Diet, Then Control Diet Alone: This group will first consume the supplement daily for 4 weeks in addition to the control diet and then cross-over to control diet alone.
  Acetylated and Butyrylated High Amylose Maize Starch: Participants will be instructed to consume HAMS-AB in two divided doses at breakfast and dinner
- Control Diet Alone, Then Supplement Intervention and Control Diet: This arm will start with the control diet alone then cross over to receive the supplement for 4 weeks in addition to the control diet.
Period: Baseline-Randomization
Arm/Group | Supplement Intervention and Control Diet, Then Control Diet Alone | Control Diet Alone, Then Supplement Intervention and Control Diet
Started | 6 | 6
Completed | 3 | 4
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 1 | 1
Period: Cross-over
Arm/Group | Supplement Intervention and Control Diet, Then Control Diet Alone | Control Diet Alone, Then Supplement Intervention and Control Diet
Started | 3 | 4
Completed | 3 | 3
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intervention Group: This arm will consume the supplement daily for 4 weeks.
  Acetylated and Butyrylated High Amylose Maize Starch: Participants will be instructed to consume HAMS-AB in two divided doses at breakfast and dinner
- Control Group: This arm will not receive the supplement for 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.98 (1.92) | 13.58 (1.07) | 14.28 (1.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 0 | 2 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 1 | 7
  Not Hispanic or Latino | 0 | 5 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in the Gut Microbiome Profile
Description: We planned to assess the effect of administering acetylated and butyrylated high amylose maize starch (HAMS-AB) on the gut microbiome profile in people with recently-diagnosed type 1 diabetes (T1D) by sequencing the gut microbiome profile.
  This measure was assesed using the absolute abundance of certain bacterial species of interest.
  The changes will be compared before and after each 4 week time period.
Time Frame: before and after completion of each 4 week sequence
Measure: Median (Inter-Quartile Range); unit: species count
Groups:
- Supplement Intervention and Control Diet: This group will consume the supplement daily for 4 weeks along with following the diabetic diet.
  Acetylated and Butyrylated High Amylose Maize Starch: Participants will be instructed to consume HAMS-AB in two divided doses at breakfast and dinner
- Control Diet Alone: This group will only follow the diabetic diet and not receive the supplement for 4 weeks.
Arm/Group | Supplement Intervention and Control Diet | Control Diet Alone
Number analyzed (Participants) | 5 | 6
species count
  Baseline Bifidobacterium Longum | 818.5 [110 to 1280] | 229 [49 to 609]
  Bifidobacteria Longum (after 4 weeks) | 1610 [382 to 1819.5] | 177 [75.5 to 924.5]
  Baseline Parabacteroides distasonis | 4964 [0 to 9782] | 2632 [1407 to 5179.5]
  Parabacteroides distasonis (after 4 weeks) | 561 [55 to 3556] | 561 [136 to 2986]

2. Secondary Outcome: Changes in the Short Chain Fatty Acid Levels in the Gut.
Description: Measurement of Short Chain Fatty Acid Levels in the Stools.
Time Frame: before and after completion of each 4 week sequence
Measure: Mean (Standard Deviation); unit: mmol / kg fecal material
Groups:
- Supplement Intervention and Control Diet: This group will consume the supplement daily for 4 weeks while following the control diet.
  Acetylated and Butyrylated High Amylose Maize Starch: Participants will be instructed to consume HAMS-AB in two divided doses at breakfast and dinner
- Control Diet Alone: This group will follow only the control diet without the supplement for 4 weeks.
Arm/Group | Supplement Intervention and Control Diet | Control Diet Alone
Number analyzed (Participants) | 5 | 7
mmol / kg fecal material
  Butyrate | 23 (6) | 19 (5)
  Propionate | 16 (9) | 16 (5)
  acetate | 60 (23) | 56 (18)

3. Secondary Outcome: Changes in Average Glucose
Description: We will compare average glucose changes pre/post intervention with HAMS-AB. We will compare their glycemic changes using continuous glucose monitoring data.
Time Frame: before and after completion of each 4 week sequence
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Control Diet Alone: This group will only follow the diabetic diet and will not receive the supplement for 4 weeks.
Arm/Group | Supplement Intervention and Control Diet | Control Diet Alone
Number analyzed (Participants) | 5 | 3
mg/dl
  baseline | 256 (19) | 228 (13)
  4 weeks after | 232 (31) | 217 (27)

4. Secondary Outcome: C-peptide Levels (Changes in Beta Cell Health).
Description: We will compare β-cell measures pre/post intervention with HAMS-AB and between the intervention and control groups. We will assess β-cell function using mixed meal tolerance-derived C-peptide measurements ( a measure of β-cell function).
Time Frame: before and after completion of each 4 week sequence
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Control Diet Alone: This group will only follow the diabetic diet for 4 weeks.
Arm/Group | Supplement Intervention and Control Diet | Control Diet Alone
Number analyzed (Participants) | 4 | 3
ng/ml
  baseline | 2.0 (0.3) | 1.7 (0.3)
  after 4 weeks | 2.7 (0.6) | 2.6 (0.4)

5. Other Pre Specified Outcome: Changes in Frequency of Mucosal Associated Invariant T (MAIT) Cells
Description: We will compare changes in MAIT cell frequency (as measured by % of CD3 T cells that are MAIT cells) before and after the interventions
Time Frame: before and after completion of each 4 week sequence
Measure: Number; unit: percentage of CD3 T cells
Arm/Group | Supplement Intervention and Control Diet | Control Diet Alone
Number analyzed (Participants) | 7 | 8
percentage of CD3 T cells
  Baseline | 2.3 | 1.6
  after 4 weeks | 2.1 | 2.4

6. Other Pre Specified Outcome: Changes in Function of Mucosal Associated Invariant T (MAIT) Cells
Description: We will compare changes in % of MAIT cell with CD25 function before and after the interventions
Time Frame: before and after completion of each 4 week sequence
Measure: Number; unit: percentage of MAIT cells
Arm/Group | Supplement Intervention and Control Diet | Control Diet Alone
Number analyzed (Participants) | 7 | 8
percentage of MAIT cells
  before | 4.7 | 3.8
  after | 3.2 | 4.0

7. Other Pre Specified Outcome: Changes in Phenotype of Mucosal Associated Invariant T (MAIT) Cells
Description: We will compare changes in % of MAIT cells with a BCL2-GzB+ phenotype before and after the interventions
Time Frame: before and after completion of each 4 week sequence
Measure: Number; unit: percentage of MAIT cells
Arm/Group | Supplement Intervention and Control Diet | Control Diet Alone
Number analyzed (Participants) | 7 | 8
percentage of MAIT cells
  before | 16.7 | 11.5
  after | 5.4 | 9.0

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: CTCAE was used for adverse and serious adverse event reporting. Data on AEs was collected at the time of each scheduled visit in addition to in between visit during phone communications.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 7/9 | 7/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention Group (N=9) | Control Group (N=10)
Dental Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
anxiety (Investigations) | 0 (0) | 1 (1)
bilateral halux infection (Infections and infestations) | 0 (0) | 1 (1)
cold (Infections and infestations) | 1 (1) | 0 (0)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
yeast infection (Infections and infestations) | 1 (1) | 0 (0)
flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
emesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)
rash at sensor insertion site (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
low vitamin D (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
sweating during blood draw (Investigations) | 0 (0) | 1 (3)
epistaxis (Vascular disorders) | 0 (0) | 1 (1)
loss of appetite (Gastrointestinal disorders) | 0 (0) | 1 (1)
CGM fell off (Product Issues) | 0 (0) | 1 (1)
Headaches (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-11): https://cdn.clinicaltrials.gov/large-docs/57/NCT04114357/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT04114357/ICF_001.pdf